CLINICAL TRIAL: NCT05844878
Title: Study Protocol for RCT of Integrative Music-mindfulness Intervention for Treating of Dental Anxiety Among Iraqi Adult Patients Seeking Private Dental Care in Karbala City.
Brief Title: Effect of Dental Anxiety Management by Integrative Music-mindfulness Intervention Among Iraqi Adult Patients in a Karbala City Private Clinic, an RCT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF CO2302/0008 (P)
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2024-07

CONDITIONS: Dental Anxiety; Behavioral Management
Keywords: dental anxiety; impact; behavioral management; adult; Iraqi patients
MeSH Terms: conditions — Tooth, Impacted | interventions — Cognitive Behavioral Therapy; Muscle Relaxation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental anxiety management intervention group (Experimental): in this arm; the patients will under go combination of 2 anxiety management techniques by using of behavioral therapeutic management including; Cognitive behavioral therapy (CBT) by using Distraction technique, and Mindfulness technique by using of relaxation breathing with muscle relaxation, during dental treatment through 30 minutes. then after 3 months those patients will be followed up for re measurement of anxiety level by using the same modified dental anxiety scale questionnaire.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) by using Distraction technique.; Behavioral: Mindfulness technique by using of relaxation breathing with muscle relaxation
- control group (No Intervention): in this arm; the patients will under go dental treatment for the same duration as the intervention arm treatment, but without applying the anxiety management techniques. Subsequently, each patient will be followed up after 3 months, similar to the intervention group.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) by using Distraction technique. — Distraction: The distraction in this arm will be done by hearing of soft music; the name of music that will be used is "relaxing piano music and water sounds 24/7 - ideal for stress relief". This music will be used in both the reception room and in the dental room treatment from the time-point that patient enters the reception room, and continues into the dental treatment room until the end of dental treatment when the patient exits the dental treatment room
  Arms: Dental anxiety management intervention group
Behavioral: Mindfulness technique by using of relaxation breathing with muscle relaxation — The mindfulness technique consist of combination of 2 procedures:
  1. Relaxation breathing: this will be done during the course of dental treatment by asking the patient to do the following "Gently breathe in - hold - and let go". This procedure will be applied at the first moment when the patient sits on the dental chair before any dental treatment is done and the patient is asked to repeat this twice, each for a duration of 10 seconds. This procedure will be repeated twice; at zero time and after an interval of 16 minutes of dental treatment that extend for a 30-minute duration for each patient.
  2. Muscle relaxation: this will be done by asking the patient during dental treatment to do the following "Hands - gently clench - hold - and let go". This procedure will be applied after 8 minutes from starting dental treatment, and ask the patient to do it twice for about 10 seconds. This procedure will be repeated twice; at 8 minutes and at 24 minutes of dental treatment.
  Arms: Dental anxiety management intervention group

SUMMARY:
Dental anxiety considered as one of the weariest problems and disturbing problems with which the individual dentist has had to fight. Dental anxiety has been a major patient's complaint which interferes with different dental treatment. Therefore, dental anxiety may have a critical impact on the deterioration of oral health. It is a problem of many patients. Excessive dental anxiety will leads to bad oral health.

It is estimated that about 36% of the world population are suffering from dental anxiety and 5- 15% of adults in developed countries suffer from severe anxiety to dental treatment. According to researchers, between 50% and 80% of adults in the United States have some degree of dental anxiety. In Saudi Arabia dental anxiety was found to be 50%. Very limited number of studies have been done in Iraq especially management of anxiety, for example in Baghdad, it was found that about 55% of study population had dental anxiety.

Because of no studies have been conducted to determine the impact of dental anxiety management in Karbala city-Iraq, thus conducting such a study is timely and much needed to improve patient care.

The goal of this clinical trial is to test the effectiveness of behavioral management technique on patients having different levels of dental anxiety, among Iraqi adult patients seeking private dental care in Karbala city.

The main question it aims to answer is: Is dental anxiety management effective in decreasing dental anxiety levels among adult Iraqi patients seeking private dental care in Karbala city? Participants will be requested to fill the self-reported questionnaire paper for anxiety levels determination & sociodemographic factors. Researchers will use non-pharmacological behavioral therapeutic techniques including combination of cognitive behavioral therapy (distraction technique) and mindfulness therapy (relaxation breathing and muscle relaxation techniques) applied as one package. the patients with anxiety will be divided in to 2 groups; one group with applying intervention and the other group without applying intervention to see if the dental anxiety therapy is effective in decreasing dental anxiety level for anxiety patient.

This study hypothesized that there is a significant difference in the changes of dental anxiety level between managed patients and not managed patients (between group) and (within group) between pre and post managed patients after three months follow up assessment.

DETAILED DESCRIPTION:
Study design:

This study is a non-pharmacological parallel randomized control trial study design (RCT). It includes a self-administered questionnaire modified dental anxiety scale (MDAS: modified dental anxiety scale), socio demographic factors questionnaire, which are filled by the patients for identifying eligible participants which is done in the first visit to the private dental clinic. Then after collection of all patients data, randomized allocation of the participants will be done to the patients with different levels of anxiety (low, moderate, and high level) into two groups; intervention group (cognitive behavioral therapy CBT & Mind fullness management which are applied as one package) and control group (without intervention) with allocation ratio of 1:1 for each level to each group.

After three months from the application of the dental anxiety management, these two groups of patients will be asked to come to the same clinic. In addition, they will be requested to fill the Modified Dental Anxiety Scale (MDAS) form again before any dental treatment. These steps will be applied to determine if there are any differences in their dental anxiety levels pre and post application of intervention and to assess if the intervention management is successful for this period. Furthermore, researchers will see the effect of management techniques on patients with and without systemic diseases and compare between them to see if there are any significant differences of the intervention on patients with and without systemic diseases. This is because some patients do not seek dental care due to anxiety from complications of systemic diseases and not due to anxiety from dental treatment procedures.

Participants:

The participants for this study design consists of Iraqi adult patients, aged 25year and above, of both genders, who have self-reported as having dental anxiety, seeking Iraqi private dental care in Karbala city for various treatment modalities with using of dental anesthesia injection, who attending private dental clinic which is located in an area named "Hay Al-amel" in the center of Karbala city.

How participants and clinic recruited to this study? This study will be applied in one private dental clinics. This private dental clinic is recruited to this study by providing all requirement needed for this study as the following;

1. This clinic consist of a reception room, dental treatment room, and third room suitable for patients' interview.
2. This clinic will provide all necessary copies of; participant information sheet (PIS), consent form, MDAS questionnaire papers for pre & post intervention treatment, sociodemographic questionnaire papers.
3. Provide microphone in both reception room and dental treatment room for hearing of soft music during dental anxiety management.

In this private clinic the patients will be treated by the same dentist that have a good experience for about 22 years. All those patients coming to this clinic were received by the same secretariat person.

The participant after acceptance to be part of this study by reading and assigning the consent form and PIS; will undergo and follow the following procedures which include:

1. Each participant come to dental clinic in the first visit will be requested to fill the self-reported questionnaire paper for MDAS & sociodemographic factors, before any dental treatment.
2. Dental treatment according to the patients need.
3. After completing data collection of all participants, then inviting the anxiety patients recruited with different levels of dental anxiety for next treatment appointment (as a second visit appointment) in the same private dental clinic by the same dentist for applying dental treatment for both arms and applying the intervention for intervention arm. The date of this visit should be recorded and fixed specifically for each patient.
4. Researchers will be going to use RCT study design to investigate the efficacy of the combination of cognitive behavioral therapy and mindfulness intervention which applied as one package for managing dental anxiety.
5. Then; each patient within the intervention arm and within the control arm will be invited for dental treatment (as a third visit appointment) and follow up after three months specifically for each patient from the date that recorded in previous patient's visit. All those patients in this visit will be recruited and invited to this visit to the same private dental clinic and treated by the same dentist. All those patients will be requested by the same secretariat person to fill a new MDAS questionnaire paper in the reception room before any dental treatment (this is the second MDAS questionnaire paper that should be filled by the same patients). Hence in this visit it is very important that those patients should be come for this visit for completing dental treatment or new dental treatment and not only for follow up to fill the MDAS questioner paper, to prevent any bias. Because the psychology and feeling of the patients are not the same when the patient go to the dentist clinic for dental treatment or go to the dentist clinic to fill MDAS questionnaire paper without any dental treatment.

Intervention: dental anxiety management (CBT & Mindfulness technique):

Researchers will be going to use (RCT) to investigate the efficacy of the combination of CBT and mindfulness intervention for managing dental anxiety. This combination intervention technique is described in the following sections.

1. CBT which include:

1. Distraction: is one of the useful techniques of diverting the patient's attention from what may be perceived as an unpleasant procedure. This enables decreased perception of unpleasantness and averting negative or avoidance behavior. The distraction in this study will be done by hearing of soft music; the name of music that will be used is "relaxing piano music and water sounds 24/7 - ideal for stress relief". This music will be used in both the reception room and in the dental room treatment from the time-point that patient enters the reception room, and continues into the dental treatment room until the end of dental treatment when the patient exits the dental treatment room.

   2. Mindfulness technique:
2. Diaphragmatic or relaxation breathing: Diaphragmatic or relaxation breathing in this study will be done during the course of dental treatment by asking the patient to do the following "Gently breathe in - hold - and let go". This procedure will be applied at the first moment when the patient sits on the dental chair before any dental treatment is done and the patient is asked to repeat this twice, each for a duration of 10 seconds. This relaxation breathing procedure will be repeated twice; at zero time of treatment and after an interval of 16 minutes of dental treatment that extend for a 30-minute duration for each patient. (That mean applied at 0 minute, then at 16 minutes).
3. Progressive muscle relaxation: The Progressive muscle relaxation in this study will done by asking the patient during dental treatment to do the following "Hands - gently clench - hold - and let go". This procedure will be applied after 8 minutes from starting dental treatment (which mean after 8 minutes from applying the relaxation breathing technique), and ask the patient to do it twice for about 10 seconds. All these procedures will be repeated twice; at 8 minutes of treatment and at 24 minutes of dental treatment that extend for a duration of 30 minutes for each patient. (That means it is applied at the 8 minute, then at the 24 minute)

The anxiety management intervention and treatment procedure used in this study will be applied for 30 minutes for each dentally anxious patient. This is done for standardization purpose. Follow up dental appointments for these patients will be after three months.

In the control group, Researchers will carry out dental treatment for the same duration as the intervention arm treatment, but without applying the anxiety management techniques. Subsequently, each patient will be followed up after 3 months, similar to the intervention group.

ELIGIBILITY:
Inclusion Criteria: Researchers will include patients who fulfill these criteria:

* All patients with self-reported anxiety score MDAS from (6 - 25) in phase one.
* All patients who are scheduled to undergo dental treatment with a planned maximum treatment length of 30 minutes are eligible to participate in the study.
* Patients accept to undergo management technique for their dental anxiety.

Exclusion Criteria: Researchers will exclude the following patients:

* Patients who have systemic diseases other than diabetes, hypertension, heart problem, and hyperthyroidism.
* Patients that did not complete the MDAS questionnaire.
* Patients that did not attend any follow up.
* Patients that refuse to complete and follow the study requirement.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
The dental anxiety measured by using modified dental anxiety scale MDAS | Post intervention measurement of MDAS after 3 months from applying the intervention
  MDAS will be used to determine anxiety levels which will be divided as the following;
  * No anxiety = (5 point)
  * Low level of anxiety = (6 - 10 point)
  * Moderate level of anxiety = (11 - 15 point)
  * High level of anxiety = (16 - 25 point). MDAS consists of five questions where by each of question has five scores, ranging from 'not anxious', 'slightly anxious', 'fairly anxious', 'very anxious' to 'extremely anxious,' in ascending order from 1 to 5.

SECONDARY OUTCOMES:
Dental anxiety management | Post intervention measurement of MDAS after 3 months from applying the intervention.
  by using modified dental anxiety scale MDAS to determine anxiety levels which will be divided as the following;
  * Low level of anxiety = (6 - 10 point)
  * Moderate level of anxiety = (11 - 15 point)
  * High level of anxiety = (16 - 25 point). the minimum MDAS score mean less anxiety level, and if the MDAS score for the same patient is less in post intervention measurement than pre intervention measurement; that is mean the management technique is successful to decrease the anxiety level for this patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Doss, Professor, Study Chair — University of Malaya
Locations (2):
- Dental Private Clinic, Karbala, Hay Al-amel, Iraq
- UM University, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
depending at the time of study ending